CLINICAL TRIAL: NCT01204268
Title: The Neuroprotection of Sevoflurane Preconditioning on Perioperative Ischemia-reperfusion Injury During Intracranial Aneurysm Surgery
Brief Title: The Neuroprotection of Sevoflurane Preconditioning on Intracranial Aneurysm Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Responsible Party: Hailong Dong, Xijing Hospital, Fourth Military Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: APC-BRAIN-2009
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Last update posted 2010-09-20 (Estimated); Status verified 2009-08

CONDITIONS: Brain Ischemia
Keywords: cerebral ischemia; sevoflurane preconditioning; intracranial aneurysm surgery
MeSH Terms: conditions — Brain Ischemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Propofol group (No Intervention): Patients will receive the total intravenous anesthesia with propofol infusion during the surgery.
- Sevo-C group (Active Comparator): Patients will receive the anesthesia with continuous inhalation of sevoflurane.
  Interventions: Procedure: Sevo continuous inhalation
- Sevo-I group (Experimental): Sevoflurane will be given before the cerebral artery clip as a preconditioning procedure for the coming ischemia-reperfusion injury.
  Interventions: Procedure: Sev-I group

INTERVENTIONS:
Procedure: Sev-I group — Sevoflurane will be given before the cerebral artery clip as a preconditioning procedure for the coming ischemia-reperfusion injury.
  Other Names: Sevoflurane preconditioning
  Arms: Sevo-I group
Procedure: Sevo continuous inhalation — Patients will receive the anesthesia with continuous inhalation of sevoflurane.
  Arms: Sevo-C group

SUMMARY:
The current study is designed to clarify the neuroprotective effect of sevoflurane preconditioning on the patients underwent intracranial aneurysm surgery.

DETAILED DESCRIPTION:
The current study is designed to clarify the neuroprotective effect of sevoflurane preconditioning on the patients underwent intracranial aneurysm surgery. The patients with cerebral aneurysm will be recruited in current study. The sevoflurane preconditioning will be performed before the surgical procedure. The neurological injury biomarkers, such as S-100b and NSE will be detected. The neurological function and recovery will be assessed after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patient under intracranial aneurysm surgery.

Exclusion Criteria:

* Patients who refused to participate or who had a history of chemotherapy/convulsions two weeks prior to admission, stroke/cardiopulmonary resuscitation/head trauma three months prior to admission, Alzheimer's disease, amyotrophic lateral sclerosis, and prior melanoma were excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-08 (Estimated); Study Completion 2011-10 (Estimated)

PRIMARY OUTCOMES:
S-100B,NSE | 7 days

SECONDARY OUTCOMES:
Karnofsky Performance Scale,NIH stroke index, MMSE | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hailong Dong, MD, PhD, Principal Investigator — Xijing Hospital
Locations (1):
- Xijing Hospital, Xi'an, Shaanxi, China